CLINICAL TRIAL: NCT01126320
Title: Frequency of Ventilator Associated Pneumonia (VAP) in Mechanically Ventilated ICU Patients Using the AnapnoGuard System
Brief Title: Frequency of Ventilator Associated Pneumonia (VAP) in Mechanically Ventilated Patients Using the AnapnoGuard System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitech Respiration (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HST -AG -02
Record Dates: First submitted 2010-05-15; First posted 2010-05-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Ventilator Associated Pneumonia
Keywords: VAP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AnapnoGuard 100 (Experimental): Respiratory guard system during mechanical ventilation
  Interventions: Device: AnapnoGuard 100,
- Control (Active Comparator): routine mechanical ventilator
  Interventions: Device: routine mechanical ventilator

INTERVENTIONS:
Device: AnapnoGuard 100, — Respiratory guard system during mechanical ventilation with routine mechanical ventilator
  Arms: AnapnoGuard 100
Device: routine mechanical ventilator — routine mechanical ventilation
  Arms: Control

SUMMARY:
Ventilator Associated Pneumonia (VAP) is a common complication experienced by mechanically ventilated patients and within the framework of Respiratory Intensive Care Units. The AnapnoGuard system, developed by Hospitech Respiration Ltd. is a ventilation guard system that includes a number of unique characteristics. This study was designed to test the frequency VAP in mechanically ventilated ICU patients using the AnapnoGuard System.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients;
* Patient was connected to AnapnoGuard system up to six hours from intubation;
* Age - above 18.

Exclusion Criteria:

* Pneumonia;
* Aspiration Pneumonia;
* Chronic or Severe Pneumonia;
* Chronic Obstructive Pulmonary Disease (COPD) requiring permanent home-based antibiotic treatment;
* Interstitial Lung Disease (ILD);
* Post Lung Transplant State;
* Immunosuppression.
* Patients ventilated in prone position
* Patient who was ventilated 3 months prior to being enrolled in the study
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-12; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
VAP occurence | 2 years

SECONDARY OUTCOMES:
Adverse events occurence | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Bar Lavi, Dr., Principal Investigator — RAMBAM Medical Center, Haifa Israel
Locations (1):
- RAMBAM Medical Center, Haifa, Israel